CLINICAL TRIAL: NCT00828672
Title: A Randomized Phase II Study of Bevacizumab, Capecitabine and Radiation Therapy With or Without Oxaliplatin in the Preoperative Treatment of Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Bevacizumab, Capecitabine and Radiation Therapy With or Without Oxaliplatin Locally Advanced Rectal Cancer
Acronym: AXEBEAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s51104 - ML5194; 2007-007177-23 (EudraCT Number); MO19051 (Other Grant/Funding Number: UZ Leuven with support from Roche and Sanofi)
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: bevacizumab; capecitabine; radiation therapy; oxaliplatin; multimodality treatments; TME (total mesorectal excision); Axe Beam; rectal cancer; neoadjuvant; pathological complete response; postoperative complications
MeSH Terms: conditions — Rectal Neoplasms; Postoperative Complications | interventions — Oxaliplatin; Bevacizumab; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AXE (ARM 1) (Active Comparator): Oxaliplatin, Bevacizumab and Capecitabine concurrently with radiotherapy.
  Interventions: Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Capecitabine; Radiation: radiotherapy
- AX (ARM 2) (Active Comparator): Bevacizumab and Capecitabine concurrently with radiotherapy
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Radiation: radiotherapy

INTERVENTIONS:
Drug: Oxaliplatin — Administered on days 15,22,29,36 en 43; 50 mg/m2
  Other Names: Eloxatin
  Arms: AXE (ARM 1)
Drug: Bevacizumab — Administered on days 1,15,29 and 43 ; 5mg/kg
  Other Names: Avastin
Drug: Capecitabine — 825 mg/m2 ; 25 days - 5days per week, concurrent with radiotherapy
  Other Names: Xeloda
Radiation: radiotherapy — Total dose 45Gy

SUMMARY:
Phase II clinical trial, open-label, randomized, two arms, multicentre (possibly multinational). Academic, investigator initiated.

To assess the activity of bevacizumab (AvastinTM) in combination with capecitabine (XelodaTM) and radiation therapy with or without oxaliplatin (EloxatinTM) in the pre-operative treatment of locally advanced rectal cancer, followed by TME (total mesorectal excision).

DETAILED DESCRIPTION:
See Synopsis

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of rectum measurable (RECIST), locally advanced (defined by MRI - Tumour beyond mesorectal fascia (T4) or Tumour ≤ 2 mm from mesorectal fascia or T3 tumour < 5 cm from anal verge
* Patient is at least 18 years of age
* Good organ function

Exclusion Criteria:

* Evidence of distant metastases
* Contraindication for bevacizumab
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Cutsem, Prof. Dr., Principal Investigator — UZ Leuven
Locations (9):
- Belgium (9):
  - Onze Lieve Vrouwziekenhuis, Aalst
  - ZNA Middelheim, Antwerp
  - AZ St- Lucas, Bruges
  - Erasme Hospital, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - AZ Groeninge, Kortrijk
  - C.H.U. Sart-Tilman, Liège
  - Clinique Sainte Elisabeth, Namur
  - H. Hartziekenhuis, Roeselare

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-four patients were included. First patient enrolled: 22-Jun-2009. Last patient enrolled: 29-Sep-2013. Participating sites: UZ Leuven, Erasme Hospital Bruxelles, Cliniques Universitaires St-Luc Bruxelles, AZ St. Lucas Brugge, AZ Groeninge Kortrijk, CHU Sart-Tilman Liege, OLVZ Aalst, H. Hart Ziekenhuis Roeselare, Cl. Saint Elisabeth Namur
Pre-assignment Details: Target population was represented by patients with locally advanced rectal cancer (tumour beyond mesorectal fascia (T4) or tumour ≤ 2 mm from mesorectal fascia or T3 tumour < 5 cm from anal verge by MRI), histologically confirmed. Pts were screened as per incl and excl criteria per protocol. Screening failures were not recorded in the eCRF.
Period: Pre-treatment (Baseline)
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Started | 43 | 41
Completed | 43 | 41
Not Completed | 0 | 0
Period: Study Treatment
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Started | 43 | 41
Completed | 41 | 39
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Complete response, no surgery | 1 | 1
Period: Post-surgery (<30 Days)
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Started | 41 | 39
Completed | 41 | 38
Not Completed | 0 | 1
Not completed — No central review materials | 0 | 1
Period: Follow-up
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Started (Pt with compl response&no surgery and pts with no central review material and with AEs joined in FU) | 42 (Patient in Arm 1 with clinical complete response and no surgery is in follow up (joined this period)) | 41 (Patients with no central review material and with adverse event are in followup (joined this period))
Completed | 42 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AXE (ARM 1) | AX (ARM 2) | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 14 | 12 | 26
Age, Continuous [Median (Full Range); unit: years] | 61 [26 to 77] | 59 [35 to 78] | 60 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 29 | 29 | 58
ECOG PS (Performance Status) [Count of Participants; unit: Participants] — ECOG PS = 0 Fully active, able to carry on all pre-disease performance without restriction; ECOG PS = 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    ECOG PS=0 | 36 | 37 | 73
    ECOG PS=1 | 7 | 4 | 11
Distance from tumour to anal verge [Count of Participants; unit: Participants] — Distance from tumour to anal verge measured during colonoscopy (in cm).
  Participants
    <5cm | 18 | 15 | 33
    >=5cm | 13 | 15 | 28
    NA | 12 | 11 | 23
Distance to CRM [Count of Participants; unit: Participants] — Distance to CRM measured by MRI
  Participants
    0mm | 21 | 24 | 45
    <2mm | 6 | 2 | 8
    >=2mm | 9 | 10 | 19
    NA | 7 | 5 | 12
Tumour stage [Count of Participants; unit: Participants] — Tumour staging was done using clinical, radiological and pathological assessments on rectal biopsies. Tumors (T) were graded using the colon and rectum cancer staging (TNM, American Joint Committee on Cancer 7th edition) where T2 tumors are less severe then T3 tumors and T4 tumors respectively.
  Participants
    T2 (Tumor invades muscularis propria) | 2 | 2 | 4
    T3 (tumor invades into pericolorectal tissues) | 34 | 31 | 65
    T4 (tumor invades through peritoneum/other organs) | 7 | 8 | 15
Nodal stage [Count of Participants; unit: Participants] — Nodal staging was done using clinical, radiological and pathological assessments where applicable. Lymph node involvement (N) was graded using the colon and rectum cancer staging (TNM, American Joint Committee on Cancer 7th edition) where N0 is no regional lymph node involved and N1 is less severe then N2 involvement.
  Participants
    N0 (no regional lymph node metastase) | 7 | 5 | 12
    N1 (metastasis in 1-3 regional lymp nodes) | 15 | 18 | 33
    N2 (metastasis in 4 or more regional lymph nodes) | 20 | 17 | 37
    Nx (regional nodes cannot be assessed) | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response at Surgery. Overview of Complete Pathologic Responses, Good and Little Tumour Regression Rates at Surgery.
Description: Dworak tumour regression grades (TRG) were used to assess pathologic response: TRG0=no regression. TRG1=dominant tumor mass with obvious fibrosis and/or vasculopathy; TRG2=dominant fibrotic changes with few tumour cells or groups; TRG3=very few (difficult to find microscopically) tumour cells in fibrotic tissue with or without mucus substance. TRG4=no intact viable tumour cells, only fibrotic mass or presence of mucin lakes without associated malignant cells (total tumour regression). Pathologic assessments of tumour response post chemoradiotherapy as provided by investigators (read by local pathologists on operative specimens) were reviewed centrally for all pts for whom surgical materials were available (centrally reviewed set). The diagnosis of independent central reviewers primed. Pathologic complete response rates (TRG4) are reported (%). Good (TRG3 and TRG4 together) and little (TRG 0,1 and 2) tumour regression rates are summarized. For these 2 last rows, % add to 100.
Time Frame: 4 months
Population: Patients who had undertaken surgery and had pathology materials available for central review (centrally reviewed subset)
Measure: Number (95% Confidence Interval); unit: percentage of cases
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Number analyzed (Participants) | 41 | 38
percentage of cases
  Pathological complete response (Dworak TRG=4) % | 34 [19 to 49] | 11 [0 to 21]
  Good tumour regression (Dworak TRG=3-4) % | 41 [26 to 57] | 24 [10 to 38]
  Little tumour regression (Dworak TRG=0-1-2) % | 59 [43 to 74] | 76 [62 to 90]

2. Secondary Outcome: Number of Participants With Histopathologic R0 and Negative CRM Resection
Description: Histopathologic R0 resection rate was defined as margins histologically negative for tumour involvement after resection. The circumferential resection margin (CRM) is considered to be involved if microscopic tumour is present <1mm from or at the inked circumferential or radial resection margin. Data on quality of mesorectal excision were expected but not collected consistently.
Time Frame: 4 months
Population: Patient in Arm 2 that discontinued chemoradiotherapy due to major toxicity and had surgery off protocol is counted here as well
Measure: Count of Participants; unit: Participants
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Number analyzed (Participants) | 41 | 39
Participants
  Negative resection margins | 40 | 37
  Positive resection margins | 1 | 2

3. Secondary Outcome: Number of Participants With Pathologic Complete Response at Surgery. Number of Participants With Good or Little Pathological Tumour Regression at Surgery.
Description: as for outcome 1
Time Frame: 4 months
Population: Centrally reviewed subset
Measure: Count of Participants; unit: Participants
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Number analyzed (Participants) | 41 | 38
Participants
  Complete response, no tumour left Dworak TRG=4 | 14 | 4
  Good tumour regression TRG=3-4 | 17 | 9
  No or little tumour regression Dworak TRG=0-1-2 | 24 | 29

4. Secondary Outcome: Clinical Response Rate
Description: Baseline tumour measurements were performed within 4 weeks prior to treatment start (RECIST). The same methods of assessment (CT and/or MRI) were used for each measurable lesion at baseline and during follow-up.
  * Complete Response (CR) is disappearance of all clinical and radiological evidence of tumour (both target and non-target lesions).
  * Partial Response (PR) is at least a 30% decrease in the sum of LD of target lesions, taking as reference the baseline sum of tumour longest diameters (LD).
  * Stable Disease (SD) is steady state of disease. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  * Progressive Disease (PD) is at least a 20% increase in the sum of LD of measured lesions taking as references the smallest sum LD recorded since the treatment started. Appearance of new lesions constitutes PD. In exceptional circumstances, unequivocal progression of non-target lesions was considered evidence of PD.
Time Frame: 3 months
Population: Intent to treat, all registered patients
Measure: Count of Participants; unit: Participants
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Number analyzed (Participants) | 43 | 41
Participants
  CR | 3 | 5
  PR | 24 | 17
  SD | 9 | 13
  PD | 0 | 1
  NA | 7 | 5

5. Secondary Outcome: Types and Numbers of Adverse Events - General Overview
Description: Adverse events graded as per NCI CTCAE (US National Cancer Institute Common Terminology Criteria for Adverse Events) version 3.0. All Serious Adverse Events occurrences are reported and counts are summarized here; all Adverse Events (all grades) related and not related to study treatment are reported and summarized here; all severe laboratory events (hematology and biochemistry Gr 3 and higher) are reported and summarized here; all severe postoperative complications (Gr 3 and higher) occurred within the first month post surgery are reported and summarized here. See section Adverse events for details.
Time Frame: continuous up to 1 year
Population: Intent to treat
Measure: Number; unit: counts of events
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Number analyzed (Participants) | 43 | 41
counts of events
  Serious adverse events | 22 | 12
  All adverse events | 564 | 426
  Severe lab events | 27 | 16
  Post operative complications at 1 month | 14 | 9

6. Secondary Outcome: Recurrence Rates and Disease Free Survival
Description: Counts and proportions of patients experiencing recurrence of disease (local and distant).
Time Frame: up to 5 years
Population: Intent to treat (one patient lost to follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Number analyzed (Participants) | 43 | 41
Participants
  Recurred Dec 2017 | 9 | 9
  Not recurred Dec 2017 | 33 | 32
  Lost to FU | 1 | 0

7. Secondary Outcome: Death Rates and Overall Survival
Description: Counts and proportions of patients deceased (post-study).
Time Frame: up to 5 years
Population: Intent to treat in follow up (one patient in Arm 1 lost to follow up).
Measure: Count of Participants; unit: Participants
Arm/Group | AXE (ARM 1) | AX (ARM 2)
Number analyzed (Participants) | 43 | 41
Participants
  Deceased (Dec 2017) | 6 | 7
  Alive (Dec 2017) | 36 | 34
  Lost to FU | 1 | 0

ADVERSE EVENTS:
Time Frame: From signature of ICF to 30 days post surgery with follow-up for residual toxicity after this period if applicable
Description: All SAE occurences are reported and displayed below. Only Gr 3-4-5 adverse events (serious and non serious) are reported in this report.
Arm/Group | AXE (ARM 1) | AX (ARM 2)
All-Cause Mortality (participants affected / at risk) | 0/43 | 1/41
Serious Adverse Events (participants affected / at risk) | 21/43 | 12/41
Other Adverse Events (participants affected / at risk) | 18/43 | 15/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXE (ARM 1) (N=43) | AX (ARM 2) (N=41)
Lung embolism (Vascular disorders) | 0 (0) | 1 (1) — Lung embolism Gr 5 - Postoperative
Neuropathy motor (Nervous system disorders) | 0 (0) | 1 (1) — Neuropathy, motor (cranial, palate, pharynx) Gr 3 (swallowing problems) - During chemoradiotherapy
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — Seizure Gr 2 in a patient with epileptic background - During chemoradiotherapy
Fever (General disorders) | 3 (4) | 0 (0) — Fever Gr 1 - During chemoradiotherapy
Depression (Psychiatric disorders) | 0 (0) | 1 (1) — Depression Gr 3 - During chemoradiotherapy
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — Rectal haemorrhage Gr 2 following rectal biopsy. During chemoradiotherapy
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) — Diarrhea Gr 3 - During chemoradiotherapy
Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) — Fistula Gr 3 - Postoperative
Leak (Gastrointestinal disorders) | 2 (2) | 3 (3) — Anastomotic leak Gr 3; 2 in arm 1 and 3 in arm 2 - all events also SAE - Postoperative
Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) — Obstruction GI Gr 2 and Gr 3; both arm 1 Postoperative
Presacral hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) — Presacral hematoma Gr 2 - Postoperative
Febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0) — Febrile neutropenia Gr 3 - During chemoradiotherapy
Septic shock (Infections and infestations) | 1 (1) | 0 (0) — Catheter related infection Gr 4 - During chemoradiotherapy
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) — Urinary tract infection Gr 2 (1 in each arm) and 1 Urinary tract infection Gr 3 in arm 1 - During chemoradiotherapy
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) — Catheter site infection Gr 3 with positive hemocultures - Postoperative
Wound infection (Infections and infestations) | 5 (5) | 2 (2) — 5 peri-anal wound infections Gr 3 (4 in arm 1; 1 in arm 2) ; 1 wound with evisceration Gr 4 in arm 1 ; 1 Gr 5 wound infection in a patient with tumor break during surgery in arm 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXE (ARM 1) (N=43) | AX (ARM 2) (N=41)
Deep venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) — DVT Gr 3 - Postoperative
Embolism (Vascular disorders) | 0 (0) | 2 (2) — Embolism Gr 4 and embolism Gr 5 - both in arm 2
Fatigue (General disorders) | 2 (2) | 1 (1) — Fatigue Gr 3 (2 pts in arm 1 and 1 pt in arm 2 - also an SAE for this pt) - during chemoradiotherapy
Depression (Psychiatric disorders) | 0 (0) | 1 (1) — Depression Gr 3 - also an SAE - during chemoradiotherapy
Sweating (General disorders) | 1 (1) | 0 (0) — Sweating Gr 3 - Postoperative
Hypertension b (Cardiac disorders) | 1 (1) | 0 (0) — Hypertension Gr 3 - baseline
Hypertension (Cardiac disorders) | 0 (0) | 2 (2) — Hypertension Gr 3 in 2 pts in arm 2 - during chemoradiotherapy
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1) — Cardiopulmonary arrest Gr 5 - FU post EOT visit
Pain pumonary/respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) — Sore throat Gr 3 and laryngeal pain Gr 3 in one patient in arm 2 - during chemoradiotherapy
Platelet count decreased (Blood and lymphatic system disorders) | 1 (2) | 0 (0) — Platelet count decreased Gr 3 - during chemoradiotherapy
Haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Hemorrhage with surgery Gr 3
Dissiminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Disseminated Intravascular Coagulation Gr 3 - during chemoradiotherapy
Hematoma postoperative (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Hematoma Gr 3 in 1 pt in arm 2 (also SAE) - postoperative
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Hematoma Gr 3 (also an SAE) - FU post EOT visit
Neuropathy sensory (Nervous system disorders) | 1 (1) | 0 (0) — Neuropathy sensory Gr 3 - during chemoradiotherapy
Syncope (Nervous system disorders) | 1 (1) | 0 (0) — Syncope Gr 3 - during chemoradiotherapy
Neuropathy - cranial (Nervous system disorders) | 0 (0) | 1 (1) — Neuropathy -cranial Gr 3 (also an SAE) - FU post EOT visit
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Pt with baseline Meniere's disease Gr 3 (since 1999) - Baseline
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Anorexia Gr 3 - during chemoradiotherapy
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0) — Diarrhea Gr 3 in 4 pts in arm 1 (three episodes were an SAE) - during chemoradiotherapy
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Pain gastro-intestinal - anal pain Gr 3
Leak Gi (Gastrointestinal disorders) | 2 (2) | 3 (3) — Leak GI Gr 3 - postoperative
Obstruction Gi (Gastrointestinal disorders) | 2 (2) | 1 (1) — Obstruction GI Gr 3 in 2 pts in arm 1 (for 1 also an SAE) and in 1 pt in arm 2 (also an SAE) - postoperative
Pain GI (Gastrointestinal disorders) | 2 (2) | 0 (0) — Stomach pain Gr 3 and pain due to leak Gr 3 - postoperative
Discharge from the anus (Gastrointestinal disorders) | 0 (0) | 1 (1) — Purulent discharge from the anus Gr - - postoperative
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) — Ascites Gr 5 - FU post EOT visit
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) — Dysphagia Gr 3 - FU post EOT visit
Leak GU (Renal and urinary disorders) | 0 (0) | 1 (1) — Leak GU Gr 5 - postoperative
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Dermatitis associated with radiotherapy Gr 3
Pain musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Pain musculoskeletal Gr 3 - Postoperative
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Rash Gr 3 - during chemoradiotherapy
Pain muskuloskeletal Gr 3 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Pain muskuloskeletal Gr 3 - postoperative
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Hypocalcemia Gr 3 - during chemoradiotherapy
Hypokalemia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Hypokalemia Gr 3 - during chemoradiotherapy
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Hyponatremia Gr 3 - during chemoradiotherapy
Febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0) — Febrile neutropenia Gr 3 (also an SAE) - during chemoradiotherapy
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) — Catheter site infection Gr 3 (also an SAE) - during chemoradiotherapy
Sepsis (Infections and infestations) | 2 (2) | 0 (0) — Sepsis Gr 3 and septic shock Gr 4 - during chemoradiotherapy
Wound infection (Infections and infestations) | 5 (5) | 2 (2) — 5 peri-anal wound infections Gr 3 ; 1 wound infection with evisceration Gr 4 ; 1 Gr 5 wound infection in a patient with tumor break during surgery
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) — Peritonitis Gr 5 (tumor break during surgery) - part of SAE
Infection due to leak of anastomosis (Infections and infestations) | 1 (1) | 0 (0) — Infection due to leak of anastomosis Gr 3 (part of an SAE) - follow-up

LIMITATIONS AND CAVEATS:
The study was not powered to allow for formal statistical comparisons between arms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is an academic institution and not the drug market authorization holder. Participating PIs were selected from other academic institutions. Participating PIs cannot publish full or partial study results before final publication by Sponsor, but they will be nominated as co-authors based on patient accrual at each participating site. Own results can be published afterwards by participant PIs, with the agreement of the Sponsor.